CLINICAL TRIAL: NCT02000869
Title: Impact of Pre- and Post-transplant Arterial Stiffness and Central Aortic Blood Pressure on Post-kidney Transplant Cardiovascular and Allograft Outcomes
Brief Title: Impact of Arterial Stiffness and Central Aortic Blood Pressure on Kidney Transplant Outcomes
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Other Study IDs: 13.0016
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- wait-listed kidney transplant candidates

SUMMARY:
People with CKD have higher prevalence of cardiovascular disease. The mechanism behind this increased risk is complex but there is strong evidence that changes in arterial stiffness play a central role. Arterial stiffness as measured by aortic pulse wave velocity (aPWV) and augmentation index (AIx), is a surrogate marker of cardiovascular organ damage, and is signiﬁcantly associated with the future risk of clinical events. In addition, aPWV is an independent and powerful predictor of all-cause and cardiovascular mortality in patients on dialysis. Reduction of aPWV, mainly by use of an angiotensin converting enzyme (ACE)-inhibitor results in an improved survival in dialysis patients. These findings suggest that arterial stiffness is not merely a marker of arterial damage but a potentially reversible factor contributing to mortality in dialysis patients. There is strong evidence that arterial stiffness increases as glomerular filtration rate (GFR) falls. Conversely, arterial stiffness has also been established in a number of studies as a significant risk factor for CKD progression.

In addition to arterial stiffness, elevated central aortic blood pressure and central pulse pressure have been shown to increase the risk of progression of CKD to ESRD. Central blood pressure is more strongly related than standard BP measured at the brachial arteries (brachial blood pressure) to concentric left ventricular hypertrophy and carotid artery hypertrophy as well as to future cardiovascular events.

Cardiovascular disease remains the foremost cause of death post-kidney transplant. Although, successful kidney transplant has been shown to improve arterial stiffness post-transplant, we do not know to what extent the pre-transplant arterial stiffness and central aortic blood pressure and their improvement post-transplant impact the cardiovascular and allograft outcomes. In addition, it is unclear what transplant related factors are associated with improvement in arterial stiffness and central aortic blood pressure post-transplant.

The goals of our study are:

1. To determine if pre-transplant central blood pressure and aortic stiffness impact post-transplant cardiovascular and kidney allograft outcomes.
2. To determine whether the changes in central blood pressure and aortic stiffness post-transplant impact cardiovascular and kidney allograft outcomes.
3. To determine the factors associated with improved central aortic blood pressure and arterial stiffness post-transplant.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a significant public health problem in United States, particularly in southern states like Louisiana. People with CKD and end-stage renal disease (ESRD) have a poor survival compared with general population, and this is primarily due to a higher prevalence of cardiovascular disease in this population. Almost 50% of deaths in patients with CKD are attributable to cardiovascular disease. The prevalence of cardiac arrhythmias, sudden cardiac death (SCD), myocardial infarction, congestive heart failure (CHF), stroke and peripheral arterial disease is all more common in patients with CKD compared with general population.

The mechanism behind the increased cardiovascular risk in this population is complex but there is a strong evidence to suggest that changes in arterial stiffness play a central role. It is known that patients with CKD and ESRD have increased arterial and aortic stiffness. Examination of the aorta and conduit arteries from patients with CKD reveals features of arteriosclerosis, a disease of the arterial medial layer. Increased collagen content, collagen cross-linking, loss of elastin, and hyperplasia and hypertrophy of vascular smooth muscle cells results in arterial wall hypertrophy which together with medial calcification promotes increased stiffness. The causes of arteriosclerosis in CKD include hypertension due to sodium retention, oxidative stress, inflammation, production of advanced glycation end products, together with activation of the renin-angiotensin-aldosterone and sympathetic nervous systems. In addition, arterial stiffness exhibits a dynamic functional component. Endothelial dysfunction resulting from high levels of oxidative stress and uremic toxins, such as asymmetrical dimethyl arginine, contributes significantly to increased arterial stiffness. Increased arterial stiffness causes adverse morphological change in the left ventricle which is believed to be the basis for CHF, lethal arrhythmia, SCD and thrombo-embolic stroke.

Arterial stiffness as measured by aortic pulse wave velocity (aPWV) and augmentation index (AIx), is a surrogate marker of cardiovascular organ damage, and is signiﬁcantly associated with the future risk of clinical events. In addition, some studies have demonstrated that aPWV is an independent and powerful predictor of all-cause and cardiovascular mortality in patients on dialysis. Reduction of aPWV, mainly by use of an ACE-inhibitor, is associated with an improved survival in dialysis patients. These findings suggest that arterial stiffness is not merely a marker of arterial damage but a potentially reversible factor contributing to mortality in dialysis patients. There is strong cross-sectional evidence that arterial stiffness increases as glomerular filtration rate (GFR) falls. In the general population, among treated hypertensives, even minimally impaired baseline renal function (serum creatinine >90μmol/l) is associated with an increased rate of aortic stiffening. Conversely, arterial stiffness has also been established in a number of studies as a significant risk factor for CKD progression.

In addition to arterial stiffness, elevated central aortic blood pressure and central pulse pressure have been shown to increase the risk of progression of CKD to ESRD. In patients with CKD, central aortic pulse pressure also positively and independently correlate with increasing brachial pulse pressure, older age, female sex, and the presence of diabetes mellitus. Furthermore central blood pressure is more strongly related than standard BP measured at the brachial arteries (brachial blood pressure) to concentric left ventricular hypertrophy and carotid artery hypertrophy as well as to future cardiovascular events.

Kidney transplantation prolongs the survival compared with dialysis, but cardiovascular disease remains the foremost cause of death post-transplant. Although, successful kidney transplant has been shown to improve arterial stiffness post-transplant, we do not know to what extent the pre-transplant arterial stiffness and central aortic blood pressure and their improvement post-transplant impact the cardiovascular and allograft outcomes. In addition, it is unclear what transplant related factors are associated with improvement in arterial stiffness and central aortic blood pressure post-transplant.

The goals of our study are:

1. To determine if pre-transplant central blood pressure and aortic stiffness impact post-transplant cardiovascular and kidney allograft outcomes.
2. To determine whether the changes in central blood pressure and aortic stiffness post-transplant impact cardiovascular and kidney allograft outcomes.
3. To determine the factors associated with improved central aortic blood pressure and arterial stiffness post-transplant.

Clinical significance of the study:

Since, arterial stiffness is not merely a marker of arterial damage but a potentially reversible factor contributing to mortality, this study may provide us an important insight into potential factors-both reversible and irreversible associated with arterial stiffness and central aortic blood pressure as well as cardiovascular morbidity and mortality and kidney allograft outcomes post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Wait-listed kidney transplant candidates who have been on the waiting list for at least 2 years

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wait-listed kidney transplant candidates who have been on the waiting list for at least 2 years
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in central aortic blood pressure and arterial stiffness post-transplant | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Singh, MD, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- John C. McDonald Regional Transplant Center, Shreveport, Louisiana, United States